CLINICAL TRIAL: NCT05684770
Title: Evaluation of Feasibility and Impact of Remote Care in Patients With Thromboembolic Disease of Low Risk
Brief Title: Impact of Remote Care in Patients Diagnosed With Thromboembolic Disease of Low Risk
Acronym: TEVEDOM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Eure-Seine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-A00894-39; CHES N°22/02 (Other: CH Eure-Seine)
Record Dates: First submitted 2022-11-07; First posted 2023-01-13 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Thromboembolic Disease
MeSH Terms: conditions — Thromboembolism | interventions — Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 4G Tablet (Experimental)
  Interventions: Other: 4G tablet

INTERVENTIONS:
Other: 4G tablet — Participants will receive for the whole period of study a 4G tablet in order to fill questionnaires, learn information about their drugs (patient education), have a remote consultation and evaluate treatment compliance.

SUMMARY:
The goal of this clinical trial is to learn about the feasibility and impact of remote care in patients diagnosed with thromboembolic disease of low risk. The main questions it aims to answer are:

* the evaluation of feasibility of organisation between different healthcare professionals (hospital physicians, primary care physician) at 6 months and 1 year
* the evaluation of complication rate, hospitalisation related to thromboembolic disease rate, compliance to treatment rate at 6 months and 1 year Participants will receive indication of treatment according to national recommendations. Additionnally, they will receive for the length of study a 4G tablet in order to fill questionnaires, learn information about their drugs (patient education), have a remote consultation and evaluate treatment compliance.

ELIGIBILITY:
Inclusion Criteria:

* patients identified in the emergency department with a thromboembolic disease, with a deep vein thrombosis or pulmonary embolism with a low risk of mortality according to recommendations
* affiliated or beneficiary of social protection

Exclusion Criteria:

* patient having a severe obstruction syndrome, a thromboembolic disease already under treatment or a suspicion of thrombocytopenia induced by heparin
* patient with an active hemorrhage or a major risk of hemorrhage, a renal severe failure, comorbidities such as cancer, or the impossibility to organise a consultation or a patient in a non favorable medico-social context
* patient with a caval thrombosis
* patient suffering of a disease at hemorrhagic risk or neurosurgery intervention done in the last month or other surgery in the last 15 days prior to inclusion
* patient with contraindication of direct oral anticoagulants, such as bitherapy with antiplatelet agent, imidazoles, macrolides, antiretroviral treatments or an anti-phospholipid syndrome
* patient that lives in an area not covered by internet
* patient that has no primary care physician
* patient not able to understand the study (language, psychological problem) or not able to read or write
* patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants in which the evaluation of medical and patient satisfaction regarding feasibility of organisation assessed by three scales (patient scale, hospital physician scale and primary care physician scale) is satisfactory | 6 months
  Three scales were created for this study :
  * patient scale : difficulty perceived to use the tablet, added value in the use of tablet, improvement of communication with physicians
  * hospital physician scale : global satisfaction (scale from 0 to 10), perception on the follow-up of patient through tablet, improvement of communication with patients and with primary care physician
  * primary care physician scale : global satisfaction (scale from 0 to 10), perception on the follow-up of patient through tablet, improvement of communication with patients and with hospital physician

SECONDARY OUTCOMES:
Number of patients in which the evaluation of medical and patient satisfaction regarding feasibility of organisation assessed by three scales (patient scale, hospital physician scale and primary care physician scale) is satisfactory | 1 year
  Three scales were created for this study :
  * patient scale : difficulty perceived to use the tablet, added value in the use of tablet, improvement of communication with physicians
  * hospital physician scale : global satisfaction (scale from 0 to 10), perception on the follow-up of patient through tablet, improvement of communication with patients and with primary care physician
  * primary care physician scale : global satisfaction (scale from 0 to 10), perception on the follow-up of patient through tablet, improvement of communication with patients and with hospital physician
Evaluation of complication rate related to thromboembolic disease | 6 months and 1 year
Evaluation of hospitalisation rate related to thromboembolic disease | 1 year
Evaluation of treatment compliance | 6 months and 1 year
  This will be evaluated by the communication between the physician and the patient during consultation

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Eble, MD, Principal Investigator — CH Eure-Seine
Locations (1):
- Centre Hospitalier Eure-Seine, Évreux, France

IPD SHARING:
Plan to Share IPD: No